CLINICAL TRIAL: NCT05723848
Title: A Prospective Study to Evaluate the Usefulness of Electronically Captured Wearable Data to Assess Disease Activity in CIDP (Chronic Inflammatory Demyelinating Polyneuropathy) Patients Undergoing IVIG (Intravenous Immunoglobulin) Treatment.
Brief Title: Electronic Monitoring of Disease Activity in Patients With Chronic Inflammatory Demyelinating Polyneuropathy
Acronym: EMDA CIDP
Status: Completed | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Dr. med. Marc Günter Pawlitzki, Principal Investigator Marc Pawlitzki, MD, Heinrich-Heine University, Duesseldorf
Other Study IDs: 2022-1881
Record Dates: First submitted 2023-01-10; First posted 2023-02-13 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: CIDP
Keywords: Smartwatch; end of dose phenomenon; neuropathy; Polyneuropathies; Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Peripheral Nervous System Diseases; Neuromuscular Diseases; Nervous System Diseases; Polyradiculoneuropathy; Autoimmune Diseases of the Nervous System; Demyelinating Diseases; Autoimmune Diseases; Immune System Diseases
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Polyneuropathies; Peripheral Nervous System Diseases; Neuromuscular Diseases; Nervous System Diseases; Polyradiculoneuropathy; Autoimmune Diseases of the Nervous System; Demyelinating Diseases; Autoimmune Diseases; Immune System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CIDP patients: CIDP patients with ongoing standard of care IVIG treatment
  Interventions: Device: Smartwatch (Withings Scanwatch)

INTERVENTIONS:
Device: Smartwatch (Withings Scanwatch) — All-day monitoring of patients via smartwatch

SUMMARY:
This clinical, prospective study aims to evaluate the usefulness of electronically captured wearable data to assess disease activity in CIDP (chronic inflammatory demyelinating polyneuropathy) patients undergoing IVIG treatment. Close clinical monitoring will complement smartwatch-acquired data to shed light on different patient clusters and end-of-dose phenomena.

DETAILED DESCRIPTION:
CIDP is a rare chronic neurological condition that leads to a considerable patient burden. As symptoms are often challenging to monitor, finding an individually optimal treatment regimen can be challenging. Additionally, patients receiving treatment often describe individual end-of-dose-phenomena, frequently leading to uncertainty regarding treatment intervals. Digital smartwatch-based measurements could add high-frequency real-world data to the picture and thus improve the understanding of individual disease courses.

Consequently, this study aims to evaluate different digital measurements and blood-based analyses to monitor disease activity in CIDP patients treated with intravenous immunoglobulins. Firstly, digital and blood-based measures will be compared to subjective patient reports and established clinical scores. Secondly, explorative analyses will aim to understand the longitudinal disease course and fluctuations thereof.

Data captured by the used smartwatches (Withings Scanwatch) includes activity-related data (step count, minutes in certain intensity levels), basic cardiovascular measurements such as heart rate, and sleep-related data (total time asleep, sleep quality, etc.). Blood-based measurements include serum neurofilament-light-chain (sNfL), glial fibrillary acidic protein (GFAP) and proteomic data. The investigators aim is to show can show whether therapy-dependent activity patterns, such as the end-of-dose phenomenon, are reflected in the recorded data.

Optionally, the digital signatures of CIDP patients will be compared to these of healthy controls wearing the smartwatch.

Patients were recruited in Düsseldorf and Münster.

ELIGIBILITY:
Inclusion Criteria:

* IVIG treated ? (all criteria a-c must be met):

  1. Documented evidence of objective response to IVIG, with clinically meaningful improvement. Clinically meaningful improvement is defined as one of the following: ≥1-point decrease in adjusted INCAT score, ≥4 points increase in I-RODS total score, ≥3 points increase in MRC Sum score, ≥8 kilopascal improvement in mean grip strength (one hand), or an equivalent improvement based on information documented in medical records and per the PI's judgement.
  2. Must be on stable IVIG therapy, defined as no change greater than 10% in frequency or dose of immunoglobulin therapy or corticosteroids within 8 weeks prior to screening
  3. Evidence of clinically meaningful deterioration on interruption or dose reduction of IVIG therapy within 24 months prior to screening, determined by clinical examination or medical records. Clinically meaningful deterioration is defined as one of the following: ≥1-point increase in adjusted INCAT score, decrease in I-RODS total score ≥4 points, decrease in MRC Sum score ≥3, mean grip strength worsening of ≥8 kilopascals (one hand), or an equivalent deterioration based on information from medical records and at the PI's judgement.

Exclusion Criteria:

* unable to use smartwatch or/and smartphone device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CIDP patients with ongoing standard of care IVIG treatment, older or 18 years
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-07-16 (Actual)

PRIMARY OUTCOMES:
Change in Inflammatory Rasch-built Overall Disability Scale (I-RODS) | Screening + Baseline (V1), After 3 months (V2), After 6 months (V3)
  24-item scale, with each item representing a common, daily activity minimum value: 0 points, maximum value: 48 points, best result: 48 points
Change in Inflammatory Neuropathy Cause and Treatment (INCAT) disability score | Screening + Baseline (V1), After 3 months (V2), After 6 months (V3)
  minimum value: 0 points, maximum value: 10 points, best result: 0 points
Change in Grip strength | Screening + Baseline (V1), After 3 months (V2), After 6 months (V3)
Change in Medical Research Council (MRC)-Sumscore | Screening + Baseline (V1), After 3 months (V2), After 6 months (V3)
  minimum value: 0 points, maximum value: 60 points, best result: 60 points
Change in Subjective occurrence of end-of-dose phenomena/wearing off | Screening + Baseline (V1), After 3 months (V2), After 6 months (V3)
Change in Quality of life (QoL) | Screening + Baseline (V1), After 3 months (V2), After 6 months (V3)
  The Quality of Life Questionnaire (QoL) is an instrument for measuring patients' subjective quality of life in a wide range of specific areas
Change in Pittsburgh Sleep Quality Index (PSQI) | Screening + Baseline (V1), After 3 months (V2), After 6 months (V3)
Change in Blood analysis (levels of sNfl, serum proteomics) | Screening + Baseline (V1), After 3 months (V2), After 6 months (V3)
Questionnaire about smartwatch usage | After 6 months (V3)
Wearing time of smartwatch (daily) | 180 days
Longitudinal development of activity parameter: step count | 180 days
Longitudinal development of activity parameter: approximate distance traveled (meter) | 180 days
Longitudinal development of activity parameter: duration of soft activity (seconds) defined by Withings | 180 days
  Examples for soft activity:
  Sleeping, Sitting quietly, Walking slowly, Typing on a computer keyboard while seated, Watching television, Doing the dishes
Longitudinal development of activity parameter: duration of moderate activity (seconds) defined by Withings | 180 days
  Examples for moderate activity:
  Walking fast, Cleaning (vacuuming, washing windows, etc.), Playing doubles tennis or badminton, Taking a bike ride, Gardening
Longitudinal development of activity parameter: duration of intense activity (seconds) defined by Withings | 180 days
  Examples for intense activity:
  Hiking, Running, Carrying heavy loads, Riding a bike, Playing football,baseball, or tennis (singles), Playing jump rope
Longitudinal development of activity parameter: sum of all active time (seconds) | 180 days
Longitudinal development of activity parameter: approximate calories burned | 180 days
Longitudinal development of sleep parameter: time awake (seconds) | 180 days
Longitudinal development of sleep parameter: number of times user woke up | 180 days
Longitudinal development of sleep parameter: time to sleep (seconds) | 180 days
Longitudinal development of sleep parameter: total time in bed (seconds) | 180 days
Longitudinal development of sleep parameter: total time asleep (seconds) | 180 days
Longitudinal development of sleep parameter: ratio of sleep/time in bed | 180 days
Longitudinal development of sleep parameter: time spent in bed before falling asleep (seconds) | 180 days
Longitudinal development of sleep parameter: time awake after first falling asleep (seconds) | 180 days
Longitudinal development of sleep parameter: Withings Sleep score | 180 days
  Defined by Withings as follows: It measures every night's sleep and provides a score out of 100 points based on 4 key inputs:
  * Duration (total time spent sleeping)
  * Depth (part of night spent in restorative phases and deep sleep)
  * Regularity (consistency between your bed- and rise-times)
  * Interruptions (time spent awake)
Longitudinal development of cardiovascular parameter: average heartrate | 180 days
Longitudinal development of cardiovascular parameter: maximal heartrate | 180 days
Longitudinal development of cardiovascular parameter: minimum heartrate | 180 days
Longitudinal development of cardiovascular parameter: time in light heartrate zone (seconds) | 180 days
  Light heartrate zone is defined by Withings as follows: from 0% inclusive to 50% exclusive of maximum heart rate.
Longitudinal development of cardiovascular parameter: time in moderate heartrate zone (seconds) | 180 days
  Moderate heartrate zone is defined by Withings as follows: from 50% included to 70% excluded of maximal heart rate.
Longitudinal development of cardiovascular parameter: time in intense heartrate zone (seconds) | 180 days
  Intense heartrate zone is defined by Withings as follows: from 70% included to 90% excluded of maximal heart rate.
Longitudinal development of cardiovascular parameter: time in maximal heartrate zone (seconds) | 180 days
  Maximal heartrate zone is defined by Withings as follows: from 90% included to 100% included of maximal heart rate.
Number and time of Irregular 1-channel ECGs (according to Withings algorithm) | 180 days

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Medical Faculty, Heinrich-Heine-University, Düsseldorf, North Rhine-Westphalia
  - University Hospital Münster, Department of Neurology, Münster, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Masanneck L, Voth J, Huntemann N, Ozturk M, Schroeter CB, Ruck T, Meuth SG, Pawlitzki M. Introducing electronic monitoring of disease activity in patients with chronic inflammatory demyelinating polyneuropathy (EMDA CIDP): trial protocol of a proof of concept study. Neurol Res Pract. 2023 Aug 24;5(1):39. doi: 10.1186/s42466-023-00267-3. PMID 37612774